CLINICAL TRIAL: NCT06101225
Title: RCT of the Effects of a Relaxation, Guided Imagery Intervention and Socioemotional Learning on the Psychophysiological Well-being, Socioemotional Regulation, Cognitive and Academic Development of Children in School
Brief Title: Effects of a Relaxation and Guided Imagery Intervention in School Context
Acronym: MR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Autónoma de Lisboa (Other)
Collaborators: Faculdade de Psicologia, Universidade de Lisboa (Unknown); ISCTE-IUL (Unknown); ISAMB - Faculdade de Medicina da Universidade de Lisboa (Unknown); Technical University of Lisbon (Other); Universidade Católica Portuguesa (Other); Universidade Lusófona de Humanidades e Tecnologias (Other); Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Iolanda Costa Galinha, Associate Professor, Universidade Autónoma de Lisboa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MindRegulation BIAL212/22
Record Dates: First submitted 2023-10-05; First posted 2023-10-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Wellness 1; Positive and Negative Affect; Social Skills; Happiness; Self Esteem; Self-Regulation, Emotion; Anxiety; Cognitive Change; Heart Rate Variability; Stress, Psychological; Physical Activity
Keywords: Guided Imagery; Relaxation; Well-being; Socioemotional Learning; Emotional Self-regulation; Psychophysiology; Randomized controled trial
MeSH Terms: conditions — Social Skills; Emotional Regulation; Anxiety Disorders; Stress, Psychological; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The RCT design includes 3 conditions to which classes (3rd and 4th graders) will be randomly allocated: the experimental group will receive MindRegulation intervention (a) relaxation and guided imagery with Socioemotional Leaning; the alternative condition group will receive relaxation intervention (b); and the waiting list control group will be involved in the regular school activities, with no intervention (c).
  Interventions (a and b) will be held during 15 minutes in class, 3 school days per week, for 5 months. Data on all measures of the study will be collected at 4 data points: before the intervention (T0), during the intervention (TIntermediate); immediately after the intervention end (T1), and at follow-up (T2), 6 months after the intervention end, for the experimental (a) and alternative condition (b) groups. After follow-up, the waiting list control group will receive intervention (a), for 5 months, after which a post-intervention measurement will be performed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data will be collected from children by independent researchers, blinded to group allocation at the three data points: before the beginning of the intervention (T0), immediately after the intervention (T1), and at follow-up (T2). In the intermediate data collection (TInt) blindness to group allocation is not possible, because data collection will be performed during the intervention. Outcome's assessors will be blinded to group assignment in all data analysis times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RegularMente Intervention (Experimental): 1. Relaxation exercises, breathing and closing the eyes, focusing on body parts;
  2. The proposal of a guided imagery through narrated scripts, leading children through the visualization of beautiful scenarios and exposure to Social and Emotional Learning content - based on the Collaborative for Academic, Social, and Emotional Learning framework (CASEL), in three major themes: Me with myself (self-awareness and self-management); Me with the others (social-awareness and relationships skills); Me with the world (responsible decision making and social awareness);
  3. Instructions for self-regulation of body posture and the use of touch (shoulders) to support children in posture regulation.
  Interventions: Other: MindRegulation Intervention
- Relaxation (Active Comparator): Relaxation exercises, breathing and closing the eyes, focusing on body parts.
  Interventions: Other: Relaxation
- Control (Other): No intervention - regular school activities.
  Interventions: Other: Waiting List Control Group

INTERVENTIONS:
Other: MindRegulation Intervention — The intervention is developed in class for 15 minutes before learning activities, three times per week, for five months - 57 sessions. Six different scripts with socioemotional learning content (based on CASEL framework) for each of the three themes will be applied.
  Other Names: MindRegulation Intervention (condition a)
  Arms: RegularMente Intervention
Other: Relaxation — The relaxation condition will be developed in the same way as in RegularMente intervention, but without the guided imagery with SEL component. Relaxation exercises applied in class 15 minutes before learning activities, three times per week, for five months - in a total of 57 sessions.
  Other Names: Relaxation (condition b)
  Arms: Relaxation
Other: Waiting List Control Group — No Intervention.
  Other Names: Control Group (condition c)
  Arms: Control

SUMMARY:
Specific aims - To test the effects of a relaxation and guided imagery intervention with socioemotional learning content on a range of socioemotional, physiological, cognitive and academic outcomes of school-aged children, measured through self-reports, neuropsychological and physiological measures, as well as teachers and parent's reports.

DETAILED DESCRIPTION:
Background: Mental imagery has long been used in psychological therapies, but only recently has research started to provide a relevant scientific basis. Imagery interventions are inexpensive and have a body of research supporting their effectiveness on behavior change, the promotion of adaptive health outcomes, the reduction of anxiety and adherence to medical interventions in adults and children. However, literature on the relaxation and guided imagery interventions benefits for children in elementary school context is very scarce. This Randomized Controlled Trial (RCT) aims to contribute to the body of research by implementing and testing the benefits of an intervention program "MindRegulation" composed of relaxation, instructions for body posture, and guided imagery with socioemotional learning (SEL), conveying adaptive beliefs about oneself, the relationships with others and the environment.

Method: The MindRegulation intervention will be developed in the classroom for 15 minutes before learning activities, three times per week, for five months, and its effects will be measured on a range of emotional, physiologic, and cognitive outcomes. Twelve classes will be randomly distributed into three conditions: (a) relaxation and guided imagery, (b) just relaxation, and (c) waitlist control. The RCT includes four data collection times: pretest, intermediate, posttest, and a six-month follow-up. The sample comprises 240 students, third and fourth graders from elementary school, between 8 and 11 years old. The variables measured in the study are: well-being, affect, anxiety, emotional regulation, socioemotional competencies, attention and processing speed, physiologic responses of arousal, stress, and well-being, and perceived benefits of the intervention. The psychometric properties of the subjective measures show they are adequate for the study population and language, except for the self-esteem scale that will be validated to the study target population.

Discussion: Improvements on the children's well-being, socioemotional regulation, cognitive function, physiologic activity and academic performance are expected after five months of MindRegulation intervention and changes on physiologic activity are expected during each MindRegulation session. Mediation effects are expected for emotional regulation, well-being and anxiety variables, from participating in the intervention in the outcome variables such as socioemotional competence, cognitive function and academic performance. Additionally, well-being and anxiety levels at pretest are expected to moderate the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Attend the 3rd and 4th grade of the selected school (8-11 years-old)

Exclusion Criteria:

* The participant classes have benefited from the RegularMind intervention previously;
* Not being able to provide self-report due to intellectual, physical or sensory disabilities.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Global Happiness Faces Scale | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Faces Scale is a single-item measure of happiness that is reliable, valid and commonly used. This scale has only 1 item but it has seven simple drawings of faces that represent participants' response options to the question: "Overall, how do you feel?". Afterwards the participants must choose the face that best represents feelings ranging from "very unhappy" to "very happy".
Positive and Negative Affect (PANAS C) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Positive and Negative Affect will be measured using a Portuguese short version of the PANAS-C. The original scale is composed of ten positive and ten negative emotions. Children rate how often they had felt each emotion under a specific time frame (e.g., over the past 2 weeks), using a 5-point scale (from 1 = very slightly or not at all to 5 = extremely). Higher scores on positive emotions and lower scores on negative emotions are indicative of higher of higher positive emotions.
Mental Health Continuum (MHC) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Mental health will be measured by the Mental Health Continuum Short Form (MHC-SF) Portuguese version. It measures positive mental health and is comprised by 14 items organized in three sub scales: emotional well-being (EWB) (3 items; e.g., "How often have you felt happy?"), social well-being (SWB) (5 items; e.g., "How often have you felt that you belong to a community such as a social group, your school, or your neighbourhood?), and psychological well-being (PWB) (6 items; e.g., "How often have you felt that you had warm and trusting relationships with others?"). This scale also provides a flourishing and languishing mental health indicator based on these three subscales: emotional well-being, social well-being, and psychological well-being. Respondents rate the frequency of each symptom of positive mental health in the past few months on a 6-point Likert type scale (0 = never to 5 = every day). Higher scores are indicative of higher Mental Health.
Socioemotional Skills - Socioemotional Skills Questionnaire (QACSE) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  The Socioemotional Skills Questionnaire QACSE adaptation for children with 9 to 12 years old derives from de QACSE for adolescents (7th to 9th grade). This instrument consists of 39 items, answered on a four-point response scale from A "Never" to D ''Always", organized into six dimensions. Higher scores are indicative of higher levels on each dimension: Self-control; Social Awareness; Relational Skills; Social Isolation; Social Anxiety; Responsible Decision Making.
Emotional Regulation Questionnaire - Children and Adolescents (ERQ-CA) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Self-Regulation of Emotions will be measure with a Portuguese version of the emotional regulation questionnaire-children and adolescents (ERQ- CA) to assess emotional control strategies. The questionnaire comprises 10 items organized in two subscales: cognitive reappraisal (6 items; e.g., When I want to feel happier, I think about something different) and expressive suppression. Responses are given on a 5-point rating scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores are indicative of higher emotional regulation in children.
Trait Anxiety Inventory for Children (STAI-C2) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Anxiety will be measured with the Trait Anxiety Inventory for Children (STAI-C2), which measures a general proneness to anxious behavior rooted in the personality as a trait. The STAI-C2 comprises 20 items and asks the children how they generally feel, most of the days. It is a self-report inventory designed to be used with upper elementary or junior high school aged children. The answers range from 1 = almost never to 3 = often. In this study, Higher scores are indicative of higher levels of trait anxiety.
Lifespan-Self-esteem-scale - (LSE) | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Self-Esteem will be measured by the Lifespan-Self-esteem-scale that is a global self-esteem scale for individuals of 5 to 89 years old. It has 4 items (e.g., "How do you feel about yourself") and the answers are registered on a 5 point scale from 1 = "really sad" to 5= "really happy". The response options are illustrated with faces expressing the appropriate feeling (e.g., really sad = crying face). Higher scores are indicative of higher self-esteem.
Wechsler Intelligence Scale for Children (WISC-III) - Subtests: Maze, Symbol Search and Code subtests (for 8 to 11 years old). | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Cognitive function as attention, processing information speed, and working memory will be assessed through: (a) Maze, Symbol Search and Code subtests of the Wechsler Intelligence Scale for Children (WISC III). The Maze subtest analyzes the ability to anticipate and plan using visuospatial strategies in working memory, the Symbol Search subtest measures the ability of perceptual discrimination, dependent on visual attention capacity and working memory, and the Code subtest measures the ability to associate numbers with symbols, and memorizing the associations in order to complete the task as quickly as possible. Higher scores on these subscales are indicative of higher cognitive function on attention and speed processing.
D2 Test | Change from baseline to post-test (at 6 months) and to follow-up (at 12 months)
  Selective and sustained attention, information processing speed, precision, and qualitative aspects related with the performance will be measured with the D2 test. It can be administered to children from 8 years of age. Its administration lasts about 8-10 minutes. It is considered a cancellation or dam test, where the individual registers a (/) on the letters "d", from left to right, while ignoring the other stimuli, on each of the 14 lines and having 20 seconds per line. Higher scores on this test is indicative of higher cognitive function, namely attention and speed processing.
Heart Rate Variability (HRV) - Electrocardiogram | Change from baseline to Intermediate (at 3 months); Change from baseline to post-test (at 6 months); and change from baseline to follow up (at 12 months).
  Heart Rate Variability (HRV) is a physiological measure of emotional regulation and well-being and it varies as a result of relaxation interventions. HRV will be calculated from continuous HR acquisition, resorting to portable and comfortable sports arm band (BItalino by Plux), with two electrocardiogram sensors attached to the upper chest with electrodes. Register will be made in two consecutive days, in the morning, during 40 minutes.
Salivary Cortisol - Physiologic Stress | Change from baseline to post-test (at 6 months)
  Salivary Cortisol - Physiologic Stress will be assessed through diurnal salivary cortisol slope, using salivettes, a reliable noninvasive method, in a subsample of 100 children. It will be collected in two days. On day one, four samples will be collected at 9.15/30h, 12.15/30h, 14.15/30h, and bedtime, with no food ingestion, washing teeth or vigorous physical activity, half an hour before assessment). On day 2, three samples will be collected at 9.15/30h, 12.15/30h and bedtime.
Skin Conductance Level - Electrodermal Activity | Change from baseline to intermediate (at 3 months); change from baseline to post-test (at 6 months); and change from baseline to follow up (at 12 months).
  Emotional activation (arousal) - Skin Conductance Level, is a measure of fluctuations in the activity of the sympathetic nervous system, and in the emotional state. It will be measured with BItalino by Plux in a comfortable arm band, with two sensors attached with two velcro rings to two fingers of the non dominant hand. Register will be made in two consecutive days, in the morning, during 40 minutes.
Actigraphy - Accelerometry | Change from baseline to intermediate (at 3 months); change from baseline to post-test (at 6 months); and change from baseline to follow up (at 12 months).
  Physical activity will be measured with an accelerometer (BItalino by Plux) in a comfortable arm band, placed in the non dominant arm, above the elbow. Measurements will be made in two consecutive mornings, during 40 minutes.
Children's semi-structured self-reports | Immediately after the intervention.
  After the last intervention session, a session will be held to collect qualitative data on the child's perception of the benefits of the intervention.
Children's Academic evaluation reports | Change from baseline to post-test (at 6 months); and to follow up (at 12 months).
  Children's Academic achievement - the complete report on each students' academic performance by the teachers, including grades, behavior and absenteeism to classes, from the 1st, 2nd and 3rd periods.
Strengths and Difficulties Questionnaire teacher's version (SDQ) | Change from baseline to post-test (at 6 months) and to follow up (at 12 months).
  Socioemotional skills of children will be measured by the Strengths and Difficulties Questionnaire teachers version (Portuguese version). The SDQ teachers' version consists of twenty-five items, organized into five scales containing 5 items and each item has three response options on a scale (not true, rated 0 or 2; hardly true, rated 1; very true, rated 2 or 0). It has 5 subscales: emotional symptoms, behavior problems, hyperactivity, relationship problems with colleagues, and prosocial behavior. Lower scores are indicative of higher socioemotional skills of children.
Teachers semi-structured reports | Immediately after the intervention.
  Teachers will be asked to reply to two semi-structured questions about their perception of the benefits of the intervention for the childrens' well-being, socioemotional and cognitive development and in what way did it contribute to the class functioning and their work with children.
Parent's semi-structured reports | Immediately after the intervention.
  Parents will be asked to reply to one semi-structured question about their perception of the benefits of the intervention for their childrens' well-being, behavior, and development.
Strengths and Difficulties Questionnaire parents version (SDQ) | Change from baseline to post-test (at 6 months); and change from baseline to follow up (at 12 months).
  Socioemotional skills of children will be measured by the Strengths and Difficulties Questionnaire parents version (Portuguese version). Socioemotional skills of children will be measured by the Strengths and Difficulties Questionnaire teachers version (Portuguese version). The SDQ parent's version consists of twenty-five items, organized into five scales containing 5 items and each item has three response options on a scale (not true, rated 0 or 2; hardly true, rated 1; very true, rated 2 or 0). It has 5 subscales: emotional symptoms, behavior problems, hyperactivity, relationship problems with colleagues, and prosocial behavior. Lower scores are indicative of higher socioemotional skills of children.

CONTACTS AND LOCATIONS:
Overall Officials: Iolanda C. Galinha, Phd, Principal Investigator — Universidade Autónoma de Lisboa
Locations (1):
- Universidade Autónoma de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brickenkamp, R., & Zilmer, E. d2 Test of Attention (d2) [Database record]. APA PsycTests. 1998. Available from: https://doi.org/10.1037/t03299-000
- [Background] Carvalho JS, Pereira S, Marques-Pinto N, Marôco A. Psychometric properties of the Mental Health Continuum-Short Form: A study of Portuguese speaking children/youths. Journal of Child and Family Studies. 2016;25(7):2141-54.
- [Background] Coelho VA, Sousa V, Marchante M. Social and Emotional Competencies Evaluation Questionnaire-Teacher's Version: Validation of a Short Form. Psychol Rep. 2016 Aug;119(1):221-36. doi: 10.1177/0033294116656617. Epub 2016 Jun 28. PMID 27356548
- [Background] Coelho VA, Sousa V. Validação do questionário de avaliação de competências socioemocionais para alunos de 1o e 2o ciclo do ensino básico. Int J Dev Educ Psychol Rev INFAD psicol. 2020;2(1):431-40.
- [Background] de Carvalho JS, Pinto AM, Marôco J. Results of a mindfulness-based social-emotional learning program on Portuguese elementary students and teachers: A quasi-experimental study. Mindfulness (N Y) [Internet]. 2017;8(2):337-50. Available from: http://dx.doi.org/10.1007/s12671-016-0603-z.
- [Background] Dias P, Gonçalves MS-C-C. Avaliação da ansiedade e da depressão em crianças e adolescentes (STAI-C-C2, CMAS-R, FSSC-R e CDI): Estudo normativo para a população portuguesa. In: Soares AP, Araújo S, Caires S, editors. Avaliação da ansiedade e da depressão em crianças e adolescentes. 1999. p. 553-64.
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559
- [Background] Harris MA, Donnellan MB, Trzesniewski KH. The Lifespan Self-Esteem Scale: Initial Validation of a New Measure of Global Self-Esteem. J Pers Assess. 2018 Jan-Feb;100(1):84-95. doi: 10.1080/00223891.2016.1278380. Epub 2017 Feb 21. PMID 28631973
- [Background] Holder MD, Klassen A. Temperament and happiness in children. J Happiness Stud [Internet]. 2010;11(4):419-39. Available from: http://dx.doi.org/10.1007/s10902-009-9149-2.
- [Background] Keyes CL. Mental health in adolescence: is America's youth flourishing? Am J Orthopsychiatry. 2006 Jul;76(3):395-402. doi: 10.1037/0002-9432.76.3.395. PMID 16981819
- [Background] Mather M, Thayer J. How heart rate variability affects emotion regulation brain networks. Curr Opin Behav Sci. 2018 Feb;19:98-104. doi: 10.1016/j.cobeha.2017.12.017. PMID 29333483
- [Background] Spielberger CD, Edwards CD, Lushene RE, Montuori J, Platzek D. The state-trait anxiety inventory for children (preliminary manual). Palo Alto, CA: Consulting Psychologists Press; 1973.
- [Background] Wechsler D. Escala de Inteligência de Wechsler para Crianças - Terceira Edição. Lisboa: Cegoc; 2003.
- [Derived] Galinha IC, de Carvalho JLDCS, de Oliveira ACP, Arriaga P, Gaspar AD, Silva HP, Ortega V. MindRegulation-SEL: randomized controlled trial of the effects of a relaxation and guided imagery intervention with socioemotional learning on the psychological and biophysiological well-being, socioemotional development, cognitive function and academic achievement of elementary school children. Trials. 2025 Jun 3;26(1):187. doi: 10.1186/s13063-025-08899-3. PMID 40462190